CLINICAL TRIAL: NCT05693948
Title: The Efficacy of Topical Serum X Containing Arbutin and Glutathione for Skin Brightening
Brief Title: The Efficacy of Topical Serum X for Skin Brightening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UMRAMREC001-22
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Healthy
Keywords: Aesthetic; Cosmetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serum X (Experimental): Participants will used serum X twice daily for 12 weeks
  Interventions: Other: Other: Serum X

INTERVENTIONS:
Other: Other: Serum X — Serum X contain arbutin and glutathione

SUMMARY:
This study is conducted to evaluate the effectiveness of topical serum X containing arbutin and glutathione for skin brightening. The study duration is 12 weeks and the skin assessment will be carried out at baseline, week 4, 8 and week 12.The main questions this study aims to answer are:

1. The skin brightening effect of the product on facial skin.
2. To observe any adverse effect occurrence with the usage of the product.

ELIGIBILITY:
Inclusion Criteria:

* Malaysia citizen
* Male and female (age 18-30 years old)

Exclusion Criteria:

* Participant with severe acne skin condition
* Participant who is taking isotretinoin, immunocompromised patients and received laser and light treatment within the last three months
* Participant who undergo whitening or cosmetic treatments such as botox and dermal fillers within the previous six month
* Participant with a history of facial surgery such as facelift or nose reshaping
* Participant with history of allergies to any ingredient in the study product
* Participant who is pregnant or plan to get pregnant

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in skin tone from baseline and at week 4, week 8, and week 12 after usage of serum X. | Baseline and at week 4, week 8, and week 12
  Skin tone will be assessed using JANUS III skin analyzer
Adverse effect after using serum X | Week 12
  Based on adverse effect occurrence on participants that occur during study period (12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ungku Shahrin Medical Aesthetic Research & Innovation (USMARI) Centre, Petaling Jaya, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No